CLINICAL TRIAL: NCT00509808
Title: Safety and Performance Evaluation of an Electro-stimulator Mounted on an Intra-oral Removable Appliance (Saliwell GenNarino) for the Treatment of Xerostomia
Brief Title: Evaluation of an Electro-stimulator for the Treatment of Xerostomia
Acronym: GenNarino
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Saliwell Ltd. (Industry)
Collaborators: Universidad El Bosque, Bogotá (Other); Charite University, Berlin, Germany (Other); University of Zagreb (Other); McGill University (Other); Istanbul University (Other); Hebrew University of Jerusalem (Other); Universita degli Studi di Palermo (Other); Universidad Nacional Autonoma de Mexico (Other); Skane University Hospital (Other); University of Brasilia (Other); Hospital San Carlos, Madrid (Other); University of Kentucky (Other); University of Helsinki (Other); Indiana University (Other)
Responsible Party: Dr. Andy Wolff, Saliwell Ltd.
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 1-Wolff
Record Dates: First submitted 2007-07-31; First posted 2007-08-01 (Estimated); Last update posted 2010-04-06 (Estimated); Status verified 2010-04

CONDITIONS: Xerostomia
MeSH Terms: conditions — Xerostomia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- electrostimulation (Sham Comparator): Use of device for predetermined length
  Interventions: Device: Electrostimulation

INTERVENTIONS:
Device: Electrostimulation — 1. 1st month GN wearing (activated or sham mode)
  2. 2nd month wearing (opposite mode)
  3. 3rd - 5th month: activated GN wearing for 1, 5 or 10 minutes
  4. 6th - 8th month: activated GN wearing for 1, 5 or 10 minutes
  5. 9th - 11th month: activated GN wearing for 1, 5 or 10 minutes
  Other Names: GenNarino

SUMMARY:
This is a multinational trial, aimed at testing the safety and performance of a electrostimulating device ("GenNarino") to treat dry mouth, over one year. The design is as follows:

* Multi-center, double blind, sham (placebo) controlled, about 10 xerostomia patients per center
* Patients receive a GenNarino (and its remote control) that is programmed for one month sham and one month active mode (the order of which is randomly assigned), and thereafter 9 months at the active mode (divided in period of 3 months, the order of each is randomly assigned at wearing GenNarino for 1, 5 or 10 minutes at a time).

Study hypothesis: Gennarino will lead to significant symptomatic improvement

- At the clinic: monthly examinations at the first 2 months, and then every 3 months, including whole saliva collection and questionnaire; at the first visit impression taking for GenNarino preparation

DETAILED DESCRIPTION:
The clinical trial, titled "Safety and performance evaluation of an electro-stimulator mounted on an intra-oral removable appliance (GenNarino) for the treatment of xerostomia" is a prospective, randomized, double-blind, sham-controlled multi-center trial, followed by an open-label study. Study subjects are patients with xerostomia. The purpose of the trial is to test the safety and efficacy of electrostimulation using the GenNarino device.

The primary endpoint is significant symptomatic improvement, and the secondary ones, increased salivary output and event free use (no adverse side-effects). The clinical follow-up consists of periodic clinical examinations.

In this clinical trial the use of the device is compared between active vs. sham mode for one month each in a double-blind design (Stage I). Thereafter, at Stage II the xerostomia relieving effect of the active device is assessed in an open label design for additional 6 months. Clinic- and home-based questionnaires and whole saliva collections are performed.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must be at least 18 years of age.
2. The patient must have clinical symptoms of xerostomia (dry mouth) due to

   * Primary or secondary Sjögren's syndrome
   * Medication intake
   * Head and neck radiation with survival expectancy of more than one year
   * Chronic graft vs. host disease with survival expectancy of more than one year
3. Patients are requested not to take systemic sialogogues during the first 2 months of the study (when active is tested vs. sham)
4. Female patients of child bearing potential must have a negative pregnancy test within twenty-four hours of enrollment.
5. The patient must understand and consent in writing to the procedure.
6. The patient agrees to undergo all examinations and clinical evaluations planned for the study.

Exclusion Criteria:

1. Active HIV or HCV infection
2. Severe systemic disease
3. Known allergy to materials similar to be used in the investigational product
4. Known mental disease
5. Presence of depression, by positive answers to both the following questions:

   * "During the past month have you often been bothered by feeling down, depressed or hopeless?"
   * "During the past month have you often been bothered by little interest or pleasure in doing things?"
6. Patients wearing other active implants like pacemaker or defibrillator
7. Patients with poor oral hygiene
8. Patients whose oral anatomical characteristics precludes the insertion of the device
9. Patients who are unable or unwilling to cooperate with study procedures.
10. Pregnancy
11. Presence of erosive or ulcerative oral lesions, which are chronic or recurrent, such as erosive lichen planus, RAS, eryth. Candidosis, and of suspected pre-malignant or malignant lesions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2007-01; Primary Completion 2008-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Significant symptomatic improvement | 1 year

SECONDARY OUTCOMES:
1- Increased salivary output 2- Event free use (no adverse side-effects) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Andy Wolff, DMD, Study Director — Saliwell Ltd.
Locations (1):
- Helsinki University Central Hospital and University of Helsinki, Helsinki, Finland

REFERENCES:
- [Derived] Strietzel FP, Lafaurie GI, Mendoza GR, Alajbeg I, Pejda S, Vuletic L, Mantilla R, Falcao DP, Leal SC, Bezerra AC, Tran SD, Menard HA, Kimoto S, Pan S, Martin-Granizo RA, Lozano ML, Zunt SL, Krushinski CA, Melilli D, Campisi G, Paderni C, Dolce S, Yepes JF, Lindh L, Koray M, Mumcu G, Elad S, Zeevi I, Barrios BC, Lopez Sanchez RM, Beiski BZ, Wolff A, Konttinen YT. Efficacy and safety of an intraoral electrostimulation device for xerostomia relief: a multicenter, randomized trial. Arthritis Rheum. 2011 Jan;63(1):180-90. doi: 10.1002/art.27766. PMID 20882668